CLINICAL TRIAL: NCT03028376
Title: S100B and Glial Fibrillary Acidic Protein (GFAP) in Prehospital Prediction of Need for Neurosurgical Observation or Intervention in Patients Suffering Moderate Traumatic Brain Injury (TBI)
Brief Title: Biomarkers in Prehospital Prediction of Need for Neurosurgical Observation or Intervention in TBI Patients
Acronym: PreTBI II
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Central Denmark Region (Other); Aarhus University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Protokol_v3_240816_PreTBI_II
Record Dates: First submitted 2016-11-21; First posted 2017-01-23 (Estimated); Last update posted 2019-04-24 (Actual); Status verified 2018-05

CONDITIONS: Traumatic Brain INjury
Keywords: biomarker; point-of-care analysis
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Moderate TBI patients: GCS 9-13
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling — Blood sampling from peripheral venous catheter routinely inserted in trauma patients during transportation

SUMMARY:
The PreTBI II study aims to investigate the diagnostic potential of prehospital S100B and GFAP measurements in prediction of need for neurosurgical observation and/or intervention in moderate TBI patients, to rule-in high-risk patients. Ultimately to select patients who will benefit from neuro surgical expertise in specialized departments and thereby possibly better patient outcome. Hopefully also minimize treatment delay, secure optimal resource consumption and streamline patient courses by predicting the presence of neurotrauma.

Hypotheses:

1. A prehospital serum S100B level > 0,10 microgram/L and expectedly above a certain and currently unknown cut-off value indicates the need for neurosurgical observation and/or intervention in moderate TBI patients.
2. A prehospital serum GFAP level above a certain and currently unknown cut-off value can significantly predict a need for urgent neurosurgical observation and/or intervention in moderate TBI patients.
3. Biomarker dynamics between prehospital and in-hospital biomarker values of S100B and GFAP can significantly predict a need for urgent neurosurgical observation and/or intervention.
4. Biomarker dynamics between prehospital and in-hospital biomarker values of S100B and GFAP can significantly predict hospital course and outcome of patients with moderate TBI.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with Glasgow Coma Score (GCS) GCS 9-13 suffering relevant trauma and displaying relevant clinical indices compatible with TBI as evaluated by EMS staff. Patients are considered incompetent due to on-going alteration of mental state.

Exclusion Criteria:

* Patients <18 years, GCS <9, >6 hours elapsed after trauma, unknown time of trauma, multi trauma, known dementia, chronic psychosis or active central nervous system (CNS) pathology.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients (≥18 years) suffering isolated head trauma and receiving an ambulance or anaesthetist-staffed critical care team dispatched by the Prehospital Emergency Medical Services (EMS) in the Central Denmark Region.
Sampling Method: Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Sensitivity of se-S100B in relation to a binary outcome measured by a yes/no question of "need for neurosurgical observation and/or intervention" pick yes/no | in relation to event within 7 days of trauma
Specificity of se-S100B in relation to a binary outcome measured by a yes/no question of "need for neurosurgical observation and/or intervention" pick yes/no | in relation to event within 7 days of trauma
Positive predictive value of se-S100B in relation to a binary outcome measured by a yes/no question of "need for neurosurgical observation and/or intervention" pick yes/no | in relation to event within 7 days of trauma
Negative predictive value of se-S100B in relation to a binary outcome measured by a yes/no question of "need for neurosurgical observation and/or intervention" pick yes/no | in relation to event within 7 days of trauma

SECONDARY OUTCOMES:
Sensitivity of se-GFAP in relation to a binary outcome measured by a yes/no question of "need for neurosurgical observation and/or intervention" pick yes/no | in relation to event within 7 days of trauma
Specificity of se-GFAP in relation to a binary outcome measured by a yes/no question of "need for neurosurgical observation and/or intervention" pick yes/no | in relation to event within 7 days of trauma
Positive predictive value of se-GFAP in relation to a binary outcome measured by a yes/no question of "need for neurosurgical observation and/or intervention" pick yes/no | in relation to event within 7 days of trauma
Negative predictive value of se-GFAP in relation to a binary outcome measured by a yes/no question of "need for neurosurgical observation and/or intervention" pick yes/no | in relation to event within 7 days of trauma

OTHER OUTCOMES:
Sensitivity of combined se-S100B and se-GFAP in relation to a binary outcome measured by by a yes/no question of "immediate treatment <24h/deferred treatment <24h" pick immediate/deferred | in relation to event within 24 hours of trauma
Specificity of combined se-S100B and se-GFAP in relation to a binary outcome measured by by a yes/no question of "immediate treatment <24h/deferred treatment <24h" pick immediate/deferred | in relation to event within 24 hours of trauma
Positive predictive value of combined se-S100B and se-GFAP in relation to a binary outcome measured by by a yes/no question of "immediate treatment <24h/deferred treatment <24h" pick immediate/deferred | in relation to event within 24 hours of trauma
Negative predictive value of combined se-S100B and se-GFAP in relation to a binary outcome measured by by a yes/no question of "immediate treatment <24h/deferred treatment <24h" pick immediate/deferred | in relation to event within 24 hours of trauma
Biomarker dynamics between prehospital and in-hospital se-S100B values in relation to a binary outcome measured by a yes/no question of "need for neurosurgical observation and/or intervention" pick yes/no | in relation to event within 24 hours of trauma
Biomarker dynamics between prehospital and in-hospital se-GFAP values in relation to a binary outcome measured by a yes/no question of "need for neurosurgical observation and/or intervention" pick yes/no | in relation to event within 24 hours of trauma
Biomarker dynamics between prehospital and in-hospital se-S100B values in relation to a binary outcome measured by a yes/no question of "favorable neurological outcome" pick favorable/unfavorable | in relation to event within 1 year of trauma
  Neurological outcome will be evaluated by a dichotomized glasgow outcome score extended (GOSE) as "Favorable (GOSE 5-8)/Unfavorable (GOSE 1-4)
Biomarker dynamics between prehospital and in-hospital se-GFAP values in relation to a binary outcome measured by a yes/no question of "favorable neurological outcome" pick favorable/unfavorable | in relation to event within 1 year of trauma
  Neurological outcome will be evaluated by a dichotomized glasgow outcome score extended (GOSE) as "Favorable (GOSE 5-8)/Unfavorable (GOSE 1-4)
Biomarker dynamics between prehospital and in-hospital combination of se-S100B, se-GFAP and se-NSE values in relation to a binary outcome measured by a yes/no question of "favorable neurological outcome" pick favorable/unfavorable | in relation to event within 1 year of trauma

CONTACTS AND LOCATIONS:
Locations (1):
- Prehospital Emergency Medical Services, Central Denmark Region, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: No